CLINICAL TRIAL: NCT03125772
Title: A Prospective, Single Blind, Multi-center, Randomized Trial to Compare the TAXUS Element™ Coronary Stent System Against the XIENCE Prime™ Coronary Stent System in the Treatment of a Diabetic Patient PopulatiOn in India
Brief Title: Trial on Safety & Performance of TAXUS Element vs. XIENCE Prime Stent in Treatment of Coronary Lesion in Diabetics
Acronym: Tuxedo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortis Escorts Heart Institute (Other)
Collaborators: Boston Scientific Corporation (Industry); Max Neeman Medical International Ltd. (Unknown)
Responsible Party: Principal Investigator, Upendra Kaul, Executive Director and Dean Cardiology, Fortis Escorts Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tuxedo; CTRI/2011/06/001830 (Registry Identifier: Clinical Trial Registry - India)
Record Dates: First submitted 2015-09-02; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Coronary Heart Disease
Keywords: coronary artery disease; diabetes mellitus; everolimus; paclitaxel stents
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Disease; Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAXUS Element™ Paclitaxel-Eluting System (Experimental): The TAXUS® Element™ stent system is a multifunctional device providing a mechanical structure for vascular lumen support and a pharmacological agent targeted toward reducing or preventing the incidence of restenosis. The TAXUS Element™ stent is a balloon expandable, stainless steel platinum alloy stent, coated with paclitaxel in a slow-release system, pre-mounted on a high-pressure Monorail delivery catheter and is intended for use in the treatment of coronary artery disease. The pharmacological agent, paclitaxel, is incorporated into a triblock polymer matrix and applied to the surface of the stent. The polymer matrix provides controlled release of available paclitaxel. The TAXUS Element™ stent design is built upon the TAXUS Express and TAXUS Liberte design experience, but incorporates several improved stent design characteristics. The TAXUS Element™ stent also has a smaller tip profile, designed to enhance the ability to cross tighter and/or more complex lesions.
  Interventions: Device: TAXUS Element™ Paclitaxel-Eluting Stent System
- XIENCE PRIME™ ™ Everolimus-Eluting Stent System (Active Comparator): The everolimus-eluting stent (EES, manufactured and distributed by Abbott Vascular, Santa Clara, CA, as XIENCE PRIME™ ) is a balloon expandable stent manufactured from a flexible cobalt chromium alloy with a multicellular design and 0.0032-in strut thickness which is coated with a thin (7.8 μm) nonadhesive, durable, biocompatible acrylic polymer and fluorinated copolymer releasing everolimus. Everolimus [40-O-(2-hydroxyethyl)- rapamycin], a semisynthetic macrolide immunosuppressant, inhibits growth factor-stimulated cell proliferation by causing cell-cycle arrest in the late G1 stage, thereby suppressing neointimal formation. Comparative analysis in an in vivo rabbit aortoiliac model has shown more rapid endothelialization with the EES compared to SES, PES, and ZES.
  Interventions: Device: Xience PRIME Everolimus-Eluting Stent System

INTERVENTIONS:
Device: TAXUS Element™ Paclitaxel-Eluting Stent System — Texus Element is the next generation Boston Scientific paclitexel-eluting coronary sten and received DCGI approval on April 13th, 2010.
  Arms: TAXUS Element™ Paclitaxel-Eluting System
Device: Xience PRIME Everolimus-Eluting Stent System — The Everolimus-eluting stent manufactured and distributed by Abbott Vascular Santa Clara, CA, as Xience Prime.
  Arms: XIENCE PRIME™ ™ Everolimus-Eluting Stent System

SUMMARY:
The TUXEDO-India is a prospective, single blind, multi-center randomized clinical trial to assess the TAXUS Element™ in a consecutive population of diabetic patients with coronary artery disease undergoing coronary revascularization. Approximately 1,830 patients with single or multi lesion, multi vessel coronary artery or saphenous vein graft disease ranging in vessels ranging from 2.25 mm to 4.0 mm in diameter by visual estimate will be enrolled in a 1:1 randomization to TAXUS Element™ vs. XIENCE™ Prime in India at up to 50 clinical sites, to demonstrate the safety and effectiveness of TAXUS Element™ in an unrestricted population.

Procedural Endpoints:

* Device success, defined as attainment of < 30% residual stenosis of the target lesion (visual assessment) using the TAXUS Element™ or XIENCE™ Prime stent.
* Lesion success defined as attainment of < 30% residual stenosis (visual assessment) using any percutaneous method.
* Procedure success defined as lesion success without the occurrence of in-hospital MACE.
* Procedure complication rate including composite and individual angiographic occurrence of dissection ≥B, distal embolization, no reflow, slow flow, abrupt closure, or perforation.

DETAILED DESCRIPTION:
Primary Endpoint:

Composite safety endpoint of Target Vessel Failure (TVF) rate at 12 months post-index procedure:

* Cardiac Death related to target vessel
* Target Vessel Myocardial Infarction (TV-MI)
* Target Vessel Revascularization (TVR)

Secondary Endpoint:

Clinical endpoints measured at 30, 180 days, and 1 and 2 years post index procedure:

* TVF rate (primary endpoint 1 year)
* Target Vessel Revascularization (TVR) rate
* Target Lesion Revascularization (TLR)
* Composite of cardiac death or target vessel MI
* Composite of all deaths, all MI, all revascularizations
* Major Adverse Cardiac Events (MACE) which is the composite endpoint of cardiac death, all myocardial infarction, and TLR
* MI (Q-wave and non-Q-wave) rate
* Cardiac death rate
* Non-cardiac death rate
* All death rate
* Cardiac death or MI rate
* All death or MI rate
* Stent thrombosis rate (definite or probable by Academic Research Consortium [ARC] definitions)

Periprocedural endpoints:

* Technical success rate
* Clinical procedural success rate

Anti-platelet Therapy

A loading dose of either Clopidogrel (300mg, 600mg recommended), Ticlopidine (500mg), or Prasugrel (60mg) must be given to the patient prior to index procedure. Thereafter, Clopidogrel (75mg daily), Ticlopidine (250mg twice daily), Prasugrel (10mg) must be given for at least 12 months after stent implantation. If the protocol mandated (loading and or daily) dosage conflicts with local DFU, the local DFU should take precedence. Aspirin (ASA): Must be administered concomitantly with Clopidogrel, Ticlopidine or Prasugrel and then continued indefinitely

Sample Size Parameters:

The expected 12 month TVF rate for both groups is estimated to be 8.4% based on the data available from the SPIRIT IV trial. Given the non-inferiority margin (delta) of 4% with equal expected means and a one-sided 5% significance level, 824 patients in each group will provide at least 90% power to reject the null hypothesis if it is false. When allowance is made for 10% attrition, approximately 915 patients are required per each treatment group. Therefore, the necessary total sample size for the trial is 1,830 patients.

ELIGIBILITY:
Inclusion Criteria:

CI1. Patient must have a diagnosis of diabetes mellitus (Type 1 or Type 2) defined according to the American Diabetes Association as history of one of the followings :

1. Two hour plasma glucose >200 mg/dL (11.1 mmol/L) following a 75g oral glucose tolerance test
2. Random plasma glucose >200 mg/dL 3. A fasting plasma glucose level >126 mg/dL (7.0 mmol/L)

4. Elevated HbA1c level 6.5 And currently undergoing pharmacological treatment 5.Patients admitted with ACS NSTEMI and HbA1c > 7 can be included even if they were not on pharmacological treatment. CI2. Patient (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed CI3. Patient is eligible for percutaneous coronary intervention (PCI) CI4. Patient has symptomatic coronary artery disease or documented silent ischemia. CI5. Patient is willing to comply with all protocol-required follow-up evaluations.

Angiographic Inclusion Criteria (visual estimate)

AI1. Target lesion must be a de novo lesion located in a native coronary artery with a visually estimated reference vessel diameter (RVD) 2.25 mm and 4.0 mm. Treatment of up to 3 de novo target lesions is allowed with a maximum of two denovo target lesions per epicardial vessel.

AI2. Target lesion length must measure 34 mm (by visual estimate) AI3. Target lesion must be in a major coronary artery or branch with visually estimated stenosis 50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow 1. AI4. If more than one target lesion will be treated, the RVD and lesion length of each must meet the above criteria. AI5. Non-study percutaneous intervention for lesions in a target vessel (including side branches) is allowed if performed 9 months prior to the index procedure. AI6. Non study percutaneous interventions for lesions in a non target vessel are allowed in the following circumstances:

1. Unsuccessful, or complicated bare metal stent, balloon dilatation, cutting balloon, atherectomy, thrombectomy, and laser treatments are allowed if performed 30 days prior to the index procedure.
2. Drug-eluting stent treatment is permitted if performed 90 days prior to index procedure. AI7. Non study, percutaneous interventions for lesion(s) in a target vessel (including side branches) or non-target vessel are allowed if performed 9 months after the index procedure.

Exclusion Criteria:

CE1. Patient has known allergy to the study stent system or protocol-required concomitant medications (e.g., stainless steel, platinum, chromium, nickel, iron, thienopyridines, aspirin, radiographic contrast medium) that cannot be adequately pre-medicated. CE2. Patient has any other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 12 months CE3. Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or 177 μmol/l) CE4. Currently participating in another investigational drug or device study

Angiographic Exclusion Criteria (visual estimate)

AE1. Target lesion meets any of the following criteria:

* Left main location including left main ostial location
* Located within 2 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery by visual estimate
* Located within a saphenous vein graft or an arterial graft or distal to a diseased arterial or saphenous vein graft. Diseased graft defined as irregularity per angiogram and any visually estimated diameter stenosis > 20%.
* Involves a bifurcation in which the side branch 2.0 mm in diameter AND the ostium of the side branch is > 50% stenosed by visual estimate.
* Involves a side branch requiring pre-dilatation
* TIMI flow 0 (total occlusion) prior to guide wire crossing
* Excessive tortuosity proximal to or within the lesion
* Extreme angulation ( ≥90°) proximal to or within the lesion
* Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified by visual estimate
* Restenotic from previous intervention
* Thrombus, or possible thrombus, present in the target vessel AE2. Patient has an additional clinically significant lesion(s) in the target vessel for which an intervention within 9 months after the index procedure may be required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1830 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Composite safety endpoint of Target Vessel Failure (TVF) rate at 12 months post-index procedure: • Cardiac Death related to target vessel • Target Vessel Myocardial Infarction (TV-MI) • Target Vessel Revascularization (TVR) | 12 Months
  TVS is defined as any ischemia-driven revascularization of the target vessel( TVR), MI (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.

SECONDARY OUTCOMES:
Target Lesion Revascularization (TLR) TVF rate (primary endpoint 1 year) Target Vessel Revascularization rate Target Lesion Revascularization Composite of cardiac death or target vessel | Measured at 30,180 days,and 1 and 2 years post index procedure
Ischemia Driven Target Lesion Revascularization (TLR) Rate TVF rate (primary endpoint 1 year) Target Vessel Revascularization rate Target Lesion Revascularization Composite of cardiac death or target vessel | Measured at 30,180 days,and 1 and 2 years post index procedure
Target Vessel Failure (TVF) | Measured at 30,180 days,and 1 and 2 years post index procedure
Ischemia Driven Target Vessel Revascularization (TVR) | Measured at 30,180 days,and 1 and 2 years post index procedure
Target Lesion Failure Rate | Measured at 30,180 days,and 1 and 2 years post index procedure
  Target Lesion Failure Rate defined as any ischemia-driven revascularization of the target lesion (TLR), MI (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel
Myocardial Infarction(MI) rate | Measured at 30,180 days,and 1 and 2 years post index procedure
  Q-wave and Non-Q-wave, cumulative and individual
Cardiac death rate | Measured at 30,180 days,and 1 and 2 years post index procedure
Non-Cardiac death rate | Measured at 30,180 days,and 1 and 2 years post index procedure
All death or MI rate | Measured at 30,180 days,and 1 and 2 years post index procedure
All Death / MI / TVR Rate | Measured at 30,180 days,and 1 and 2 years post index procedure
Major Adverse Cardiac Event (MACE) | Measured at 30,180 days,and 1 and 2 years post index procedure
  MACE defined as a composite of death, MI (Q-wave and non-Q-wave), emergent coronary artery bypass surgery (CABG), or target lesion revascularization (TLR) by repeat PTCA, or CABG.
Stent Thrombosis Rate | Measured at 30,180 days,and 1 and 2 years post index procedure
  Stent thrombosis(ST) rate defined using ARC definition of definite and probable stent thrombosis and categorized as early, late or very late.

OTHER OUTCOMES:
Device Success | Baseline
  Device Success Defined as attainment of <30% residual stenosis of the target lesion (visual assessment) using the TAXUS Element or XIENCE Prime stent.
Lesion Success | Baseline
  Lesion success defined as attainment of <30% residual stenosis (visual assessment) uring any percutaneous method
Procedure Success | Baseline
  Procedure success defined as lesion success without the occurrence of in-hospital MACE.
Procedural complication rate | Baseline
  Procedural complication rate including composite and individual angiographic occurrence of dissection, distal embolization, no reflow, slow flow, abrupt closure, or perforation

CONTACTS AND LOCATIONS:
Overall Officials: Upendra Kaul, M.D, Principal Investigator — Fortis Escorts Heart Institute
Locations (1):
- Fortis Escorts Heart Institute, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] www.crf.org/crf/newsroom/news/news-archive/963-announcing-the-tct-2015-late-breaking-trials-and-first-report-investigations